CLINICAL TRIAL: NCT01705665
Title: Histopathology of the Aspirated Thrombus During Acute Myocardial Infarction
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: HYMC-70-10
Record Dates: First submitted 2012-10-10; First posted 2012-10-12 (Estimated); Last update posted 2012-10-23 (Estimated); Status verified 2012-10

CONDITIONS: Thrombosis; Acute Coronary Syndrome
MeSH Terms: conditions — Thrombosis; Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Aspirated Coronary Thrombi During AMI

SUMMARY:
This study was initiated on the preliminary premise that a thrombus whose formation was triggered by a thrombogenic substrate, such as within an atherosclerotic plaque (Tissue factor initiated thrombus), may evolve differently than the one evolving at the site of a recently implanted stent (foreign body triggered). Consequently, the thrombus composition of a de novo clot could differ from the other one, extracted during the occurrence of a subacute thrombosis, regarding the number of various cells, the amount of fibrin and platelet aggregates and the relationship among these components. In addition, it seems relevant to evaluate the numbers and the distribution of the local monocytes, once these cells may interact with platelets (via cell -adhesion mechanisms e.g., by CD31 [PECAM-1]) and by the extrinsic coagulation pathway (via TF/FVII elaborated by plaque-resident macrophages). Such a distinction, if eventually found, may reveal the mechanisms of thrombosis within coronary arteries, and may have clinical implications.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute coronary syndrome who undergo angiography
* Evidence of coronary thrombus
* Undergo aspiration procedure yielding thrombus fragments

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted for an acute coronary syndrome who undergo angiography, found to have a coronary thrombosis that is aspirated and which yields thrombus fragments.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2012-01; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Evaluation of Possible Difference in Composition of Thrombi Aspirated during Acute Myocardial Infarction Precipitated by de novo vs Subacute Thrombosis | two years
  Analysis of thrombotic specimen contents aspirated during Acute Myocardial Infarction by searching for possible differences in the components of the thrombotic debris, whether cellular, or fibrin and platelets, in accordance with clinical parameters.

CONTACTS AND LOCATIONS:
Locations (1):
- Heart Institute, Hillel Yaffe Medical Center, Hadera, Israel